CLINICAL TRIAL: NCT00772135
Title: Pulmonary Hypertension in Adolescents and Adults With Congenital Heart Disease
Brief Title: Reversibility by Sildenafil of Exercise-Induced Abnormal Right Ventricular Pressure Response in ASD and VSD-Operated Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: Norwegian Foundation for Health and Rehabilitation (Other); Pfizer (Industry)
Responsible Party: Steinar Johansen, Foreningen for Hjertesyke Barn
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: RH 2008 HR 2006 / 2 / 0012 TM; 2006 / 2 / 0012
Record Dates: First submitted 2008-10-14; First posted 2008-10-15 (Estimated); Last update posted 2008-10-15 (Estimated); Status verified 2008-10

CONDITIONS: Congenital Heart Disease
Keywords: pulmonary hypertension; congenital heart defects; exercise; phosphodiesterase inhibitors; Exercise induced pulmonary arterial hypertensive response in congenital heart disease
MeSH Terms: conditions — Heart Defects, Congenital; Hypertension, Pulmonary; Motor Activity | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: sildenafil citrate — capsule of 50 mg , 90 minutes before exercise study

SUMMARY:
The purpose of this study is to determine whether oral sildenafil citrate reduces the abnormal right ventricular pressure response during exercise in adolescent and adult patients with specific types of congenital heart defects.

DETAILED DESCRIPTION:
13.3 Study design and protocol

13.3.1 Design: double-blind case-control cross-over study

13.3.2 Patients inclusion / exclusion criteria:

The study consists of 12-16 patients from the main study (see main protocol) who are selected by following criteria

* Abnormal right ventricular pressure response to exercise (cut-off 45 mmHg maximal RVSP during exercise)
* Informed consent to participation including use of sildenafil / placebo. The patients will be approximately one year older than during the initial study.

13.3.3 Examination protocol

The patients will be examined similarly twice with at least 12 hours and one night sleep between these activities to ensure drug washout. One hour before each study part, a pharmacy produced capsule (envelope coded and drawn in a random manner from a box) containing either sildenafil citrate 50 mg or placebo will be administered. In this manner each patient will be tested once with placebo use and once with sildenafil use respectively.

The participant is taken to a clinical exercise physiology laboratory for testing separated by a night's sleep and at least 12 hours.

Monitoring equipment is mounted during the period of drug absorbtion and distribution.

1. One minute handgrip static exercise is performed as described with 80% of maximal strength applied. BP response is registered beat to beat.
2. Pulmonary function is examined, including pulmonary volumes (single breath, technical description see below), and spirometry
3. Cardiopulmonary exercise testing according to main protocol (see 3.8)
4. Exercise echocardiography during supine bicycle exercise is performed as described in main protocol (see 3.7). Other monitoring during supine cycle exercise:

   1. ECG
   2. Diffusion capacity is monitored (intra breath, technical description below). For equipment calibration haemoglobin concentration is measured by fingertip blood sampling before and after cycle exercise.
   3. Cardiac output and peripheral oxygen saturation is continuously monitored by Task Force Monitor (see below)
5. Pulmonary function testing is repeated
6. Handgrip testing is repeated as in 1.

Difffusion capacity monitoring There are two ways of measuring diffusion capacity using SensorMedics V-max analyzing system (Yorba Linda, CA, USA) - intra breath and single breath.

Measurements of forced vital capacity (FVC), forced expiratory volume (FEV1), FEV1 ratio (FEV1/FVC), peak expiratory flow (PEF), total lung capacity (TLC or VA), diffusion capacity for carbon monoxide (TLCO), adjusted diffusing capacity (TLCO/VA), residual volume (RV), capillary blood volume (Vc) and membrane conductance (Dm) are included in the analysis and will be performed according to European Respiratory Society standards.

Single breath The diffusion capacity is used to estimate the amount of gas travelling from lungs to the bloodstream across the membrane. In the process methane (CH4) is used in the concentration of 0.3 %, 0.3 % carbon monoxide (CO), 21 % oxygen (O2) and nitrogen (N2). In the estimation of TLCO several measurements are included; 1) the area of gas transportation between alveoli and the capillaries (A), 2) the wall thickness (membrane) between the alveoli and the erythrocytes (T), 3) the amount of haemoglobin available (Hb) and 4) the reaction rate of CO too Hb (θ) are determinants for the amount of CO that manage to diffuse across to the blood57.

In the process CH4 is used as a marker, as it does not diffuse across to the blood but become diluted. CH4 mixes with the residual volume in the lungs, and the degree of dilution is used to calculate alveoli volume. CO diffuses across to the blood in addition to become diluted. By measuring the amount of CO and CH4 in the expiration air compared to the inhaled gas, after a hold of breath in 8-10 seconds, we get an expression for the diffusion capacity in the lungs.

Figure 1: The single-breath method for TLCO Intra breath Intra breath reefers to the continuous real-time measurement of carbon monoxide uptake by the pulmonary capillary blood during a single breath maneuver. Intra breath maneuver may be performed during exercise.

The calibration procedure samples to set the span points to 0.3 % CO and 0.3 % CH4 (methane). The patient starts with normal breathing and is then instructed to exhale as much as possible - then inhale completely. After total inhalation the patient should exhale at a slow even flow until the computer end the test. The test window shows gas concentration versus time and volume versus time tracing in real time during the maneuver. The flow versus time curve is shown simultaneously. The collection interval used in the calculation of the TLCO is extending from 20 - 80 % of the exhaled volume (marked area in figure 2).

Figure 2. The intra breath method for TLCO

The patients need to practice this maneuver at rest before using it during exercise. The exhalation time is reduced during exercise, but the patients must try to exhale as slowly as they can in order for the analysis to be correct.

Cardiopulmonary monitoring and analysis When analysing changes in vascular resistances during exercise a measurement of pressure is only a part of the hemodynamic picture. According to Ohms law, blood flow measurement is necessary to conclude about the vascular resistances. For this purpose, a non-invasive cardiac stroke volume analyser based on thoracic impedance technique, will be used.(Task Force Monitor, CNS systems, product description enclosed) This equipment is validated for cardiac output monitoring as compared with thermodilution as gold standard. Combined with a beat to beat finger cuff system for measurement of blood pressure, this machine produces core circulatory parameters continuously. Autonomic nervous function (BP variation, HR variation) and baroreflex sensitivity is also analysed.

Continuous measurement of peripheral oxygen saturation is registered with Masimo SET pulse oximeters.

13.4 Statistics

Responses with and without sildenafil will be compared within same individual. For parameters affected by calibration differences in machinery from test 1 to 2 delta values will be compared.

Power analysis:

Data from the main study allow estimations of anticipated results and statistical power. If the average of maximal RVSP during exercise in our group is 50 mmHg and sildenafil causes a 20% decrease in average to 40 mmHg (SD 10.0) a sample size of 13 patients leads to statistical power of 81.7% with 5% confidence level (calculation: DSS research 10.7.2008, http://www.dssresearch.com/toolkit/spcalc/power_a2.asp

ELIGIBILITY:
Inclusion Criteria:

* Exercise right ventricular systolic pressure of 45 mm Hg or above.
* Operated for atrial septal defect or ventricular septal defect or minimal defect not operated or minimal residual defect.

Exclusion Criteria:

* Acute infectious/febrile illness,
* Significant mental or physical disability preventing reliable exercise testing

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-02 (Estimated); Study Completion 2009-04 (Estimated)

PRIMARY OUTCOMES:
Right ventricular pressure as measured by max velocity of tricuspid valve regurgitation | baseline and max exercise

SECONDARY OUTCOMES:
DLco (lung diffusion test) | baseline and max exercise
cardiac output | baseline and max exercise

CONTACTS AND LOCATIONS:
Locations (1):
- Rikshospitalet University Hospital, Oslo, Oslo County, Norway